CLINICAL TRIAL: NCT03004053
Title: Feasibility Testing of a Novel Endoscope for Reflectance Confocal Microscopy of Normal Oral Tissue In Vivo
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-1652
Record Dates: First submitted 2016-12-21; First posted 2016-12-28 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Oral Tissue
Keywords: Reflectance Confocal Microscopy; Normal Oral Tissue; 16-1652
MeSH Terms: interventions — Endoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Volunteers will be identified by the Head and Neck Service: 25 volunteers (Part I - 8 volunteers. Part II - 17 volunteers). during the course of 12 months. The volunteers will be imaged with the endoscope, and the images will be evaluated visually and with qualitative (descriptive) statistics.
  Interventions: Device: Reflectance Confocal Microscopy (RCM) endoscope device

INTERVENTIONS:
Device: Reflectance Confocal Microscopy (RCM) endoscope device

SUMMARY:
The purpose of this study is to obtain images (pictures) of normal oral tissue, which occur inside the mouth, using a special camera. These pictures will be used in our research to evaluate a new technology that uses a laser and takes pictures of the microscopic structure of tissue. The technology is called "reflectance confocal microscopy."

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Ability to sign informed consent
* Age ≥ 18 years.

Exclusion Criteria:

* Inability to give informed consent.
* Previously known oral disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Head and Neck clinic
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
number of images with acceptable quality | 1 year
  Each image will be scored either 1 (completely unacceptable), 2 (unacceptable), 3 (possibly acceptable), 4 (acceptable) or 5 (very acceptable) relative to a reference standard The reference standard for appearance of adequate sectioning, resolution and contrast and for detectability of nuclear and cellular features will be the appearance of images and image quality, which we are intimately familiar with, based on the past several years of experience with the existing RCM device for which images of oral mucosa have been well-characterized, well-correlated to histology, and thus are well-understood.

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Patel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm